CLINICAL TRIAL: NCT00789594
Title: Improving Laboratory Monitoring in Community Practices: A Randomized Trial
Acronym: LabMon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Simon, Principal Investigator, VA Boston Healthcare System
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: R18HS017201-01 (AHRQ); R18HS017201-01 (AHRQ)
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Monitoring; Testing; Medications; Patients receiving medications and having laboratory tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Laboratory Monitoring (Experimental): Laboratory Monitoring
  Interventions: Behavioral: laboratory monitoring alerts
- Result management (Experimental): Result management
  Interventions: Behavioral: Result management module
- Both interventions (Experimental): Both laboratory monitoring and result management interventions
  Interventions: Behavioral: laboratory monitoring alerts; Behavioral: Result management module
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: laboratory monitoring alerts — laboratory monitoring alerts
  Arms: Both interventions; Laboratory Monitoring
Behavioral: Result management module — Result management module
  Arms: Both interventions; Result management

SUMMARY:
The investigators propose a cluster-randomized controlled trial (RCT) of computerized point-of-care alerts in the EHR to prevent errors related to laboratory monitoring at the initiation and continuation of drug therapy and a results management system to prevent errors related to the delay in follow-up of abnormal laboratory testing.

DETAILED DESCRIPTION:
Medication errors and preventable adverse drug events occur commonly among patients in the ambulatory setting and constitute an important target for patient safety and quality improvement. Laboratory monitoring to ensure the safety and effectiveness of drug therapy and the timely management of abnormal results of laboratory testing have been increasingly recognized as important areas for improving patient safety in ambulatory care. Promising interventions have been developed for practices affiliated with hospitals and integrated delivery systems, but efforts to date have not adequately reached physicians practicing solo or in small practices in the community. The Massachusetts e-Health Collaborative (MAeHC; www.maehc.org) provides an important opportunity to study implementation of healthcare information technology innovations in a community setting. In 2007, the MAeHC will complete the implementation of commercially available electronic health records (EHRs) for 441 physicians in more than 200 office practices in three diverse communities in Massachusetts. In this group of small-to-medium sized office practices in both urban and rural regions of the State, we will: 1) identify the barriers to and facilitators of laboratory monitoring and timely follow-up of abnormal laboratory results, especially for elderly patients and clinical scenarios common to this population; 2) design, implement and evaluate the effectiveness of clinical decision support (point-of-care alerts) for laboratory monitoring in a widely used, commercially available EHR; 3) design, implement and evaluate the effectiveness of a results management system to improve the timely follow-up of abnormal laboratory test results in office practice; 4) develop a practical dissemination guide to assist other practices and communities interested in implementing similar interventions. The results of this study will be important because they will demonstrate and accelerate the dissemination of clinicians' use of healthcare information technology to improve patient safety and healthcare quality beyond integrated delivery systems and should be broadly generalizable to small- and medium-sized office practices in community settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care from clinicians at primary care and adult internal medicine specialty practices

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Laboratory Monitoring | 6-months

SECONDARY OUTCOMES:
Result management | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Simon, MD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States